CLINICAL TRIAL: NCT03225014
Title: A Pilot Study in the Management of Adolescent Anterior Knee Pain: Electromyostimulation Compared to Standard Physical Therapy
Brief Title: Adolescent Anterior Knee Pain: ARP Wave Therapy vs. Physical Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rady Children's Hospital, San Diego (Other)
Collaborators: STACK Velocity San Diego (Unknown)
Responsible Party: Principal Investigator, Eric Edmonds, Orthopedic Surgeon, Rady Children's Hospital, San Diego
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 151837
Record Dates: First submitted 2017-02-16; First posted 2017-07-21 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Knee Pain Chronic

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Physical Therapy (Active Comparator)
  Interventions: Diagnostic Test: Physical therapy
- ARP Wave Therapy (Active Comparator)
  Interventions: Device: Accelerated Recovery Performance Wave Therapy

INTERVENTIONS:
Device: Accelerated Recovery Performance Wave Therapy — ARP Wave therapy utilizes direct current compounded with a high frequency double exponential background waveform that creates an electromyostimulation with characteristics that contrast with more conventional therapeutic neuromuscular electrical stimulation, including: interferential, microcurrent, galvanic, Russian stimulation, and iontophoresis. ARPWave therapy is a class II FDA medical device that has been approved for muscle re-education, relaxation of muscle spasms, increased neovascularization, prevention of disuse atrophy, and maintaining/increasing joint range of motion. The ARPWave Rx100 uses a main electrostimulation pulse of 40 to 500 cycles per second that is coupled with a background high-frequency carrier signal at 10,000 cycles per second. The polarity direction of electron flow is reversible within the unit and this is utilized as part of the therapy.
  Other Names: ARP Wave therapy
  Arms: ARP Wave Therapy
Diagnostic Test: Physical therapy — PT protocol for traumatic knee pain focuses on flexibility and development of hip core strength over a 6 week period, visiting the therapist twice per week and encouraged to maintain a home exercise program (HEP). They will all receive a handout with basic exercises to use at home to ensure that progress with their HEP is maximized (Appendix I). Basic stretches for the hamstring and quadriceps muscles will also be provided with line drawings. During this treatment period the patients will complete a daily diary of time spent on the HEP with attestation from their parents or guardians, in order to improve compliance.
  Other Names: PT
  Arms: Physical Therapy

SUMMARY:
Accelerated Recovery Performance (ARP) Wave therapy is an electromyostimulation therapy designed to enhance neuromuscular control in order to rehabilitate patients with musculoskeletal pathology. The outcomes of this technology have not been assessed under the rigors of clinical science. This prospective randomized crossover study will assess ARP Wave to both shorten duration of therapy and determine other advantages in the treatment of adolescent anterior knee pain. Two cohorts of teenagers will be followed weekly through either physical therapy (PT) or ARP Wave therapy, physiological therapy versus neurological therapy, respectively. Results should highlight the clinical utility of this modality and provide pilot data for future study.

DETAILED DESCRIPTION:
This study will utilize a prospective randomized cohort of adolescent patients that present to the orthopedic sports center (age restriction greater than 12 years old) with adolescent anterior knee pain. This knee pain includes: Osgood-Schlatter disease, Sindig-Larsen-Johanssen syndrome, patellofemoral syndrome, symptomatic medial plicae, and Hoffa fat pad syndrome/impingement. Although these diagnoses affect slightly different sites at the anterior knee, the underlying pathology is essentially the same: muscle inflexibility and core strength weakness. These are clinical diagnoses, and plain radiographs are expected to be normal with no significant osseous abnormalities other than possible apophyseal fragmentation. Skeletal maturity will not be an exclusion criteria; but, previous surgery, history of hemarthrosis, previous physical therapy due to lack of control within the cohorts, and/or diagnosis of ligament, meniscal, cartilage, or tendon injury will be criteria for exclusion.

Randomization by computer generated order of consent packets will be utilized once the family and patient agrees to undergo treatment via the proposed trial. Two cohorts of patients will be created: Cohort #1 and #2. Cohort #1 will consist of patients that begin with the PT portion of the study (2 sessions per week for 6 weeks per standard of care) and cross-over in the ARP Wave protocol (20 sessions over 4 weeks). Cohort #2 will consist of patients that begin with the ARP Wave protocol and then cross-over in the standard PT protocol.

Both cohorts will undergo physical therapy utilizing a standard of care uniform PT protocol for a traumatic knee pain that focuses on flexibility and development of hip core strength over a 6 week period, visiting the therapist twice per week and encouraged to maintain a home exercise program (HEP). They will all receive a handout with basic exercises to use at home to ensure that progress with their HEP is maximized (Appendix I). Basic stretches for the hamstring and quadriceps muscles will also be provided with line drawings. During this treatment period the patients will complete a daily diary of time spent on the HEP with attestation from their parents or guardians, in order to improve compliance.

Both cohorts will undergo the same ARP Wave protocol, as well. There are 20 sessions that are used to take a single individual through to completion of treatment over a period of 30 days. During that time frame the athletes are not allowed to undergo PT, HEP or their normal athletic endeavors since it may interfere with the neuromuscular training particular to this therapeutic modality. Treatments will be performed at an outside vendor that has agreed to perform the treatments at reduced cost for the sake of this study.

Both cohorts of patients will be evaluated every two weeks, for 10 weeks, by an independent team of observers who will be blinded to the actual cohort that the patient is randomized. These individuals will perform a Return to Sports (RTS) assessment and measurement of thigh circumference of the patients at these biweekly assessments. Although the RTS will not provide an objective measure of absolute core muscle strength, it does provide an objective measure of dynamic muscle function - which is the ultimate objective of these treatment modalities, not absolute strength of any given muscle such as the quadriceps. Moreover, the RTS makes an objective assessment of both strength and endurance of the core lower extremity muscle groups. These independent observers will also administer patient-derived outcome scores.

An interim analysis for each patient will be performed once they complete their first arm of the study. Both the research staff and the orthopedic surgeon principal investigator (PI) will examine the outcome variables at this time in insure safety in treatment. If the patients are scoring in the 95% percentile on all outcome measures, they will be considered as reaching the study endpoint and will not cross-over into the next phase of treatment. For patients who do not reach this 95% percentile of healing at the end of the first arm, crossover into the next arm of the study will occur immediately. At the end of 10 weeks and successful completion of both arms of the study, the patient will be seen by the orthopedic surgeon to make a final assessment regarding treatment progress, knee pain, and whether or not further treatment will be required (in the standard of care for these patients, regardless of study cohort).

ELIGIBILITY:
Inclusion Criteria:

* Osgood-Schlatter disease, Sindig-Larsen-Johanssen syndrome, patellofemoral syndrome, symptomatic medial plicae, and Hoffa fat pad syndrome/impingement

Exclusion Criteria:

* Previous knee surgery
* History of hemarthrosis
* Previous physical therapy (PT)
* Diagnosis of ligament, meniscal, cartilage, or tendon injury.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01-09 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Return to Sport test | through study completion, an average of 10 weeks
  objective assessment of both strength and endurance of the core lower extremity muscle groups

SECONDARY OUTCOMES:
Pedi-IKDC outcome score | through study completion, an average of 10 weeks
  assesses knee function in adolescents and children
Kujala outcome score | through study completion, an average of 10 weeks
  assesses knee function in adolescents and children
Marx outcome score | through study completion, an average of 10 weeks
  assesses knee function in adolescents and children

CONTACTS AND LOCATIONS:
Locations (1):
- Rady Children's Hospital, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Only those personnel listed on the IRB-approved study protocol will have access to IPD.